CLINICAL TRIAL: NCT06197256
Title: Right and Left Ventricular Dysfunction in Critically Ill COVID-19 Patients and the Effects of Inhaled Nitric Oxide: A Sub-study of a Prospective Randomized Controlled Trial
Brief Title: Cardiac Dysfunction in Critically Ill Covid-19 Patients
Status: Completed | Type: Observational
Sponsor: Region Stockholm (Other Government)
Collaborators: Karolinska Institutet (Other)
Responsible Party: Sponsor
Other Study IDs: iNO Cardiac
Record Dates: First submitted 2024-01-08; First posted 2024-01-09 (Actual); Last update posted 2024-01-09 (Actual); Status verified 2024-01

CONDITIONS: COVID-19; ARDS, Human; Cardiac Failure; Right Ventricular Dysfunction; Left Ventricular Dysfunction; Pulmonary Hypertension
MeSH Terms: conditions — COVID-19; Respiratory Distress Syndrome; Heart Failure; Ventricular Dysfunction, Right; Ventricular Dysfunction, Left; Hypertension, Pulmonary

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
We conducted an observation sub-study of the prospective randomized controlled trial "High Dose Inhaled Nitric Oxide in Acute Hypoxemic Respiratory Failure", in which we analysed the echocardiographic data collected both at baseline when patients where included and 3-5 days later for followup.

DETAILED DESCRIPTION:
We conducted an observation sub-study of the prospective randomized controlled trial "High Dose Inhaled Nitric Oxide in Acute Hypoxemic Respiratory Failure" which was conducted in 2020/2021 during the COVID-19 pandemic on patients with ARDS due to COVID and requiring mechanical ventialtion. Patients underwent echocardiography at baseline, and were then randomized either to control, or treatment with inhaled nitric oxide, starting at 80ppm and then 40ppm. Followup echocardiography was performed 3-5 days later, and all echocardiographies were conducted by highly experienced sonographeres certified by the European Association of Cardiovascular Imaging. Analysis of these cardiac ultrasounds focused on the amount of patients showing signs of pulmonary hypertension, right ventricular failure and left ventricular failure. Several parameters were used to estimate these, and we also aimed to evalute the utility of more novel measures such as RV and LV GLS for this use in the ICU.

ELIGIBILITY:
Inclusion Criteria:

* Age ≥18.
* Positive PCR for COVID-19.
* Admission to the ICU.
* Endotracheal intubation and mechanical ventilation.
* Severe hypoxemia, defined by PaO2/FiO2 < 300 mmHg.
* Inclusion in the trial "High Dose Inhaled Nitric Oxide in Acute Hypoxemic Respiratory Failure"

Exclusion Criteria:

* Endotracheal intubation for >72h before inclusion.
* Do not resuscitate order or other limitation of care.
* Known pregnancy.
* Cases where the treating physician opposes inclusion due to safety concerns or considerations that renders inclusion unfeasible.
* Not having had echocardiography performed during the trial period (exclusion criteria for this sub-study).

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: A population studied in the trial "High Dose Inhaled Nitric Oxide in Acute Hypoxemic Respiratory Failure", consisting of 40 patients recruited in the ICU at Danderyds Hospital at the height of the COVID-19 pandemic. The study population consisted of critically ill patients requiring mechanical ventilation suffering from verified COVID-19 with ARDS.
Sampling Method: Probability Sample
Enrollment: 39 (Actual)
Dates: Start 2020-05-07 (Actual); Primary Completion 2021-02-11 (Actual); Study Completion 2021-02-11 (Actual)

PRIMARY OUTCOMES:
Delta MPAP | 3-5 days
  Difference in MPAP, measured at baseline and at followup
Delta RV GLS | 3-5 days
  Difference in RV GLS, measured at baseline and at followup
Delta TAPSE | 3-5 days
  Difference in TAPSE, measured at baseline and at followup

SECONDARY OUTCOMES:
Delta EF | 3-5 days
  Difference in EF, measured at baseline and at followup
Delta CI | 3-5 days
  Difference in CI, measured at baseline and at followup
Delta LV GLS | 3-5 days
  Difference in LV GLS, measured at baseline and at followup
Rates of LV failure detected by LV GLS compared to EF | Presented both at baseline and followup
  Comparison of the amount of patients with LV failure for LV GLS and for EF, presented at both timepoints
Rates of RV failure detected by RV GLS compared to TAPSE | Presented both at baseline and followup
  Comparison of the amount of patients with RV failure for RV GLS and for TAPSE, presented at both timepoints
Associations between levels of pulmonary hypertension, PEEP, peak pressures, central venous pressures and measurements | 3-5 days
  Regression analysis will be performed to check for association between these potential confounders

OTHER OUTCOMES:
Associations between levels of pulmonary hypertension, PEEP, peak pressures, central venous pressures and measurements | Baseline and followup 3-5 days later
  Regression analysis will be performed to check for association between these potential confounders and RV function, to be corrected for if applicable

CONTACTS AND LOCATIONS:
Overall Officials: Daniel Törnberg, MD PhD, Study Director — KI DS
Locations (1):
- Danderyds Hospital, Stockholm, Sweden

IPD SHARING:
Plan to Share IPD: No